CLINICAL TRIAL: NCT01870102
Title: A Randomized, Open Label, Cross-over, Phase 1 Trial to Investigate the Pharmacokinetics in Multi-dose and the Food Effect in Single-dose of Pelubiprofen IR and Pelubiprofen SR in Healthy Male Volunteers
Brief Title: Phase 1 Study to Compare the Pharmacokinetic Characteristics and Food Effect of Pelubiprofen (30mg) Tablet IR and Pelubiprofen SR (as a Pelubiprofen 45 mg) Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DW330SR-1002(Ver1.1.)
Record Dates: First submitted 2013-06-03; First posted 2013-06-05 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Males
MeSH Terms: interventions — pelubiprofen; BID protein, human

ARMS (4):
- Pelubiprofen IR (Pelubiprofen 30 mg) (Active Comparator)
  Interventions: Drug: Pelubiprofen IR (Pelubiprofen 30mg) TID
- Pelubiprofen SR (Pelubiprofen 45 mg) (Experimental)
  Interventions: Drug: Pelubiprofen SR (Pelubiprofen 45 mg) BID
- Pelubiprofen SR (Pelubiprofen 45 mg) fasting condition (Other)
  Interventions: Drug: Pelubiprofen SR (Pelubiprofen 45 mg) BID
- Pelubiprofen SR (Pelubiprofen 45 mg) fed condition (Other)
  Interventions: Drug: Pelubiprofen SR (Pelubiprofen 45 mg) BID

INTERVENTIONS:
Drug: Pelubiprofen IR (Pelubiprofen 30mg) TID
  Arms: Pelubiprofen IR (Pelubiprofen 30 mg)
Drug: Pelubiprofen SR (Pelubiprofen 45 mg) BID
  Arms: Pelubiprofen SR (Pelubiprofen 45 mg); Pelubiprofen SR (Pelubiprofen 45 mg) fasting condition; Pelubiprofen SR (Pelubiprofen 45 mg) fed condition

SUMMARY:
Part 1 : A randomized, open Label, multiple doses, cross-over, phase I trial to investigate the pharmacokinetics of Pelubiprofen IR (Pelubiprofen 30mg) TID and Pelubiprofen SR (Pelubiprofen 45 mg) BID in healthy male volunteers Part 2 : A randomized, open label, single dose, cross-over, Phase I trial to investigate the food effect of Pelubiprofen SR (Pelubiprofen 45 mg) in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy males aged 20~40 years
* BMI valued over 19 kg/m2, below 27 kg/m2
* Subjects whose blood pressure ; systolic BP over 90mmHg below 140mmHg, diastolic BP over 60mmHg below 90mmHg, stable station pulse over 45 bpm below 100 bpm
* Subjects who agree with double protective contraception or able to certificate already sterilization operation 1 day before administration of Investigational new drugs within 14 days after completion
* Subjects who voluntarily agreed with written consent

Exclusion Criteria:

* Subjects with clinically significant disease or past medical history in hepatic, renal, GI tract, respiratory, musculoskeletal, endocrine, neuropsychiatry, blood tumor and cardiovascular system
* Subjects with GI tract disease (eg. Crohn's disease, peptic ulcer etc.) or surgery (except appendectomy and herniotomy) influence on administration Investigational new drugs
* Subjects with hypersensitivity reaction or clinically significant disease in drugs (Aspirin, NSAID anti-inflammatory agents and antibiotics) including Pelubiprofen and Food

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
(Part1) Cmax,ss of Pelubiprofen IR (Pelubiprofen 30mg) | 0(pre-dose), 0.25h, 0.5.h, 0.75h, 1h, 1.5h, 2h, 4h, 6h, 6.5h, 7h, 8h, 12h, 12.5h, 13h, 14h, 24h, 60h, 72h, 72.25h, 72.5h, 72.75h, 73h, 73.5h, 74h, 76h, 78h, 80h, 84h, 96h (total 30 times)
(Part1) Cmax,ss of Pelubiprofen SR (Pelubiprofen 45 mg) | 0(pre-dose), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 13h, 14h, 16h, 24h, 60h, 72h, 72.5h, 73h, 73.5h, 74h, 74,5h. 75h. 75.5h, 76h, 77h, 78h, 80h, 84h, 96h (total 32 times)
(Part1) Dose normalized AUCτ,ss of Pelubiprofen IR (Pelubiprofen 30mg) | 0(pre-dose), 0.25h, 0.5.h, 0.75h, 1h, 1.5h, 2h, 4h, 6h, 6.5h, 7h, 8h, 12h, 12.5h, 13h, 14h, 24h, 60h, 72h, 72.25h, 72.5h, 72.75h, 73h, 73.5h, 74h, 76h, 78h, 80h, 84h, 96h (total 30 times)
(Part1) Dose normalized AUCτ,ss of Pelubiprofen SR (Pelubiprofen 45 mg) | 0(pre-dose), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 13h, 14h, 16h, 24h, 60h, 72h, 72.5h, 73h, 73.5h, 74h, 74,5h. 75h. 75.5h, 76h, 77h, 78h, 80h, 84h, 96h (total 32 times)
(Part2) Cmax of Pelubiprofen IR (Pelubiprofen 30mg) | 0(pre-dose), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 10h, 12h, 24h (15times each period, total 30 times)
(Part2) Cmax of Pelubiprofen SR (Pelubiprofen 45 mg) | 0(pre-dose), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 10h, 12h, 24h (15times each period, total 30 times)
(Part2) AUClast of Pelubiprofen IR (Pelubiprofen 30mg) | 0(pre-dose), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 10h, 12h, 24h (15times each period, total 30 times)
(Part2) AUClast of Pelubiprofen SR (Pelubiprofen 45 mg) | 0(pre-dose), 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 10h, 12h, 24h (15times each period, total 30 times)